CLINICAL TRIAL: NCT03431337
Title: Treatment of Acute Sinusitis With High-Dose vs. Standard-Dose Amoxicillin/Clavulanate: A Confirmation Study
Brief Title: Treatment of Acute Sinusitis With High-Dose vs. Standard-Dose Amoxicillin/Clavulanate
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Futility found by interim analysis
Sponsor: Paul Sorum, MD (Other)
Responsible Party: Sponsor-Investigator, Paul Sorum, MD, Professor of Internal Medicine and Pediatrics, Albany Medical College
Organization: Albany Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4993
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Sinusitis, Acute
MeSH Terms: conditions — Sinusitis | interventions — Amoxicillin; Lactase

STUDY DESIGN:
Intervention Model Description: 1. Ill adult patients coming to a primary care office will be diagnosed by the treating physicians with acute bacterial sinusitis in accordance with the guidelines of the Infectious Disease Society of America.
  2. If they do not meet exclusion criteria, they will be offered enrollment in the study.
  3. If they agree, they will be provided unlabeled study medication, either amoxicillin/clavulanate 875/125 + placebo pills bid x 7 days (standard dose) or amoxicillin/clavulanate 875/125 + amoxicillin immediate-release 875 (high dose).
  4. Outcomes will be assessed, by telephone or over the web (through Qualtrics), at 3 and 10 days after enrollment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unlabeled bottles of study medications, identified only by participant #, prepared by the pharmacist member of research team. The placebo will be similar in appearance to plain amoxicillin. The pills inside the bottle will be difficult to see until the bottle is opened by the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose (Experimental): Amoxicillin/clavulanate 875mg/125mg & amoxicillin 875 mg twice a day x 7 days
  Interventions: Drug: Amoxicillin 875 mg
- Standard dose (Active Comparator): Amoxicillin/clavulanate 875 mg/125mg & placebo (lactase) twice a day x 7 days.
  Interventions: Dietary Supplement: Placebo (lactase)

INTERVENTIONS:
Drug: Amoxicillin 875 mg — Doubling the dose of amoxicillin by adding amoxicillin 875 to each dose of the standard treatment of amoxicillin/clavulanate 875/125
  Other Names: Amoxil
  Arms: High dose
Dietary Supplement: Placebo (lactase) — Placebo (in place of additional amoxicillin in experimental arm)
  Arms: Standard dose

SUMMARY:
Comparative-effectiveness study of the treatment of acute bacterial sinusitis with amoxicillin/clavulanate 875mg/125mg bid for 7 days with or without the addition of immediate-release amoxicillin 875 mg bid x 7 days. .

DETAILED DESCRIPTION:
Double-blind comparative-effectiveness study of the treatment of acute bacterial sinusitis with standard dose of amoxicillin/clavulanate 875mg/125mg bid for 7 days, as recommended by the Infectious Disease Society of America, with or without the addition of immediate-release amoxicillin 875 mg bid x 7 days. The study aims are 1) to confirm, or not, our recent findings of more rapid improvement in overall symptoms with the additional amoxicillin, but also of more frequent diarrhea and vaginal yeast infections and 2) to assess, from the participants' point of view, the balance between improvement and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 and older who are patients at the Albany Medical Center Internal Medicine and Pediatrics practice (study site).
2. Clinical diagnosis of acute bacterial sinusitis in accordance with the guidelines of the Infectious Disease Society of America (fitting into one of 3 categories: persistent sinus symptoms for 10 days or more; severe sinus symptoms for 3 days or more; or worsening sinus symptoms after initial improvement (double sickening).

Exclusion Criteria:

1. Previous enrollment in the current study
2. Allergy or intolerance to any penicillin or to amoxicillin/clavulanate
3. Serious hypersensitivity reaction to any beta lactam
4. Elevated risk of amoxicillin-resistant bacteria: a. amoxicillin, penicillin, or other beta-lactam within the past month; b. known to have had methicillin-resistant Staph aureus
5. Chronic or recurrent "sinus" problems (defined as a) persistent symptoms of "sinus" congestion, not attributed to nasal allergies, for 8 weeks or more or b) 2 or more episodes of antibiotic-treated "sinusitis" in past 3 months
6. Need to use high-dose amoxicillin/clavulanate or levofloxacin or to send to emergency department or to hospitalize because of a) signs of severe infection or b) immunocompromise
7. Cognitive impairment, so unable to give reliable symptom ratings (even if a health proxy can give consent)
8. Pregnant women and nursing mothers
9. Drug warnings: a) taking allopurinol; b) current mononucleosis; c) chronic kidney disease stage 4 (estimated glomerular filtration rate <30); d) hepatic impairment (not including isolated transaminase elevated < 2 times upper limit of normal); e) history of antibiotic-associated colitis (C. difficile)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul C Sorum, MD, PhD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center Internal Medicine and Pediatrics, Cohoes, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be made available to other researchers by contacting the corresponding author at sorump@amc.edu.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately and indefinitely
Access Criteria: Contact the corresponding author at sorump@amc.edu

REFERENCES:
- [Background] Chow AW, Benninger MS, Brook I, Brozek JL, Goldstein EJ, Hicks LA, Pankey GA, Seleznick M, Volturo G, Wald ER, File TM Jr; Infectious Diseases Society of America. IDSA clinical practice guideline for acute bacterial rhinosinusitis in children and adults. Clin Infect Dis. 2012 Apr;54(8):e72-e112. doi: 10.1093/cid/cir1043. Epub 2012 Mar 20. PMID 22438350
- [Background] Lemiengre MB, van Driel ML, Merenstein D, Young J, De Sutter AI. Antibiotics for clinically diagnosed acute rhinosinusitis in adults. Cochrane Database Syst Rev. 2012 Oct 17;10:CD006089. doi: 10.1002/14651858.CD006089.pub4. PMID 23076918
- [Background] Canafax DM, Yuan Z, Chonmaitree T, Deka K, Russlie HQ, Giebink GS. Amoxicillin middle ear fluid penetration and pharmacokinetics in children with acute otitis media. Pediatr Infect Dis J. 1998 Feb;17(2):149-56. doi: 10.1097/00006454-199802000-00014. PMID 9493813
- [Background] Wald ER, Nash D, Eickhoff J. Effectiveness of amoxicillin/clavulanate potassium in the treatment of acute bacterial sinusitis in children. Pediatrics. 2009 Jul;124(1):9-15. doi: 10.1542/peds.2008-2902. PMID 19564277
- [Derived] Gregory J, Huynh B, Tayler B, Korgaonkar-Cherala C, Garrison G, Ata A, Sorum P. High-Dose vs Standard-Dose Amoxicillin Plus Clavulanate for Adults With Acute Sinusitis: A Randomized Clinical Trial. JAMA Netw Open. 2021 Mar 1;4(3):e212713. doi: 10.1001/jamanetworkopen.2021.2713. PMID 33755168

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose | Standard Dose
Started | 78 | 79
Completed | 49 | 57
Not Completed | 29 | 22
Not completed — Lost to Follow-up | 21 | 19
Not completed — Withdrawal by Subject | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- High Dose: Amoxicillin 875 mg/clavulanate 125 mg + amoxicillin 875 mg twice a day x 7 days
- Standard Dose: Amoxicillin 875 mg/clavulanate 125 mg + placebo
- Total: Total of all reporting groups
Arm/Group | High Dose | Standard Dose | Total
Number analyzed (Participants) | 78 | 79 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (15.8) | 48.5 (16.2) | 48.5 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 60 | 117
  Male | 21 | 19 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Smoking (No. [%] [Count of Participants; unit: Participants] | 12 | 7 | 19
Asthma or COPD [Count of Participants; unit: Participants] | 13 | 7 | 20
Diabetes [Count of Participants; unit: Participants] | 4 | 6 | 10
Allergic rhinitis [Count of Participants; unit: Participants] | 10 | 21 | 31
Heart disease [Count of Participants; unit: Participants] | 3 | 3 | 6
History of sinusitis [Count of Participants; unit: Participants] | 19 | 22 | 41
Hospitalized in past month [Count of Participants; unit: Participants] | 0 | 0 | 0
Antibiotics in past month [Count of Participants; unit: Participants] | 1 | 3 | 4
Using nasal steroids [Count of Participants; unit: Participants] | 18 | 19 | 37
Enrolled in previous study [Count of Participants; unit: Participants] | 10 | 7 | 17
Days of illness prior to enrollment [Mean (Standard Deviation); unit: days] | 13.9 (6.0) | 17.1 (11.0) | 15.4 (8.9)
Sinusitis category 1 (duration 10 days or greater) [Count of Participants; unit: Participants] | 54 | 58 | 112
Sinusitis category 2 (severe symptoms) [Count of Participants; unit: Participants] | 5 | 6 | 11
Sinusitis category 3 (double sickening) [Count of Participants; unit: Participants] | 18 | 12 | 30
Sinonasal Outcome Test-16 total score [Mean (Standard Deviation); unit: units on a scale] — Sum of the ratings of 16 symptoms of illness on the scale of 0 (no problem) to 3 (severe problem), with a possible range of 0 to 48, with a higher sum indicating more troubling symptoms.
  units on a scale | 29.4 (7.4) | 29.4 (8.0) | 29.4 (7.7)
Tend to be constipated [Count of Participants; unit: Participants] | 15 | 19 | 34
Prone to diarrhea [Count of Participants; unit: Participants] | 11 | 16 | 27
Tend to get vaginal yeast infections [Count of Participants; unit: Participants] | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Global Rating of Improvement of 5 & 6 at the End of 3 Days of Treatment
Description: Rating on a scale of 1=a lot worse, 2=a little worse, 3=the same, 4=a little better, 5=a lot better, 6=no symptoms, with a higher score indicating greater improvement.
Time Frame: At end of 3 days of treatment
Population: Participants who provided a Global Rating of Improvement when contacted at the end of 3 days of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Standard Dose
Number analyzed (Participants) | 66 | 70
Participants | 24 | 31

2. Secondary Outcome: Number of Participants With a Global Rating of Improvement of 5 or 6 at End of 10 Days Since Enrollment
Description: Rating of 5 (a lot better) or 6 (no symptoms) on Global Rating of Improvement scale, with range of 1 (a lot worse) to 6 (no symptoms), with a higher score indicating greater improvement
Time Frame: At end of 10 days since enrollment
Population: Participants who could be reached to give a global rating at the end of 10 days since enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Standard Dose
Number analyzed (Participants) | 49 | 57
Participants | 35 | 47

3. Secondary Outcome: Change From Baseline in the Total Score on the Sinonasal Outcome Test-16 (SNOT-16) at the End of 3 Days of Treatment
Description: The change between enrollment and the end of 3 days of treatment in the total score on the Sinonasal Outcome Test-16 (SNOT-16). The total SNOT-16 is the sum of the participant's ratings of 16 symptoms of illness on the scale of 0 (no problem) to 3 (severe problem), with a possible range of 0 to 48, with a higher sum indicating more troubling symptoms. A decrease in total score would indicate an improvement in symptoms.
Time Frame: At end of 3 days of treatment
Population: Participants who provided a SNOT-16 rating when reached at the end of 3 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose | Standard Dose
Number analyzed (Participants) | 65 | 71
score on a scale | 13.3 (8.8) | 12.3 (11.5)

4. Secondary Outcome: Change From Baseline in the Total Score on the Sinonasal Outcome Test-16 (SNOT-16) at the End of 10 Days Since Enrollment
Description: The change between enrollment and the end of 10 days since enrollment in the total score on the Sinonasal Outcome Test-16 (SNOT-16). The total SNOT-16 is the sum of the participant's ratings of 16 symptoms of illness on the scale of 0 (no problem) to 3 (severe problem), with a possible range of 0 to 48, with a higher sum indicating more troubling symptoms. A decrease in total score would indicate an improvement in symptoms.
Time Frame: At end of 10 days since enrollment
Population: Participants who could be reached at 10 days since enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose | Standard Dose
Number analyzed (Participants) | 49 | 56
score on a scale | 18.4 (11.4) | 21.4 (10.2)

5. Secondary Outcome: Balance of Benefits and Detriments
Description: Assessment of balance between good effects and bad effects of antibiotic on scale of -3=bad effects much greater than good effects to +3=good effects much greater than bad effects
Time Frame: At end of 10 days since enrollment
Population: Participants who could be reached to assess their treatment at 10 days since enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose | Standard Dose
Number analyzed (Participants) | 48 | 58
score on a scale | 1.8 (1.8) | 2.2 (1.5)

6. Secondary Outcome: Number of Participants Answering "Yes" to Willingness to Take the Antibiotic Again in the Future
Description: Response of "yes" at the end of 10 days since enrollment to the question whether the participant would take this antibiotic again, with possible answers of yes, no, or uncertain.
Time Frame: At end of 10 days since enrollment
Population: Participants who could be reached at day 10 to assess their treatment
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Standard Dose
Number analyzed (Participants) | 48 | 58
Participants | 34 | 47

7. Other Pre Specified Outcome: Number of Participants Reporting Any Diarrhea at Day 3 Among Those Self-identified as Prone or Not Prone to Diarrhea
Description: Among those who indicated at enrollment whether prone to diarrhea or not, the number giving ratings of 1, 2, or 3 on diarrhea scale ranging from 0 (none) to 3 (severe)
Time Frame: At the end of 3 days
Population: Participants giving a rating of diarrhea at the end of day 3
Measure: Count of Participants; unit: Participants
Groups:
- Prone to Diarrhea: Answering yes to baseline question of whether prone to diarrhea
- Not Prone to Diarrhea: Answering no to baseline question of whether prone to diarrhea
Arm/Group | Prone to Diarrhea | Not Prone to Diarrhea
Number analyzed (Participants) | 26 | 105
Participants | 16 | 41

8. Other Pre Specified Outcome: Number of Participants Reporting Severe Diarrhea at Day 3 Among Those Self-identified as Prone or Not Prone to Diarrhea
Description: Among those reporting proneness to diarrhea or not at enrollment, the number rating 3 on diarrhea scale ranging from 0 (none) to 3 (severe)
Time Frame: At end of day 3
Population: Participants who indicated whether prone to diarrhea or not at enrollment and then at follow-up rated their diarrhea
Measure: Count of Participants; unit: Participants
Arm/Group | Prone to Diarrhea | Not Prone to Diarrhea
Number analyzed (Participants) | 26 | 105
Participants | 4 | 6

9. Other Pre Specified Outcome: Number of Participants Reporting Any Diarrhea at Day 10 Among Those Self-identified as Prone or Not Prone to Diarrhea
Description: Among those indicating at enrollment a proneness or not to diarrhea, the number giving ratings of 1, 2, or 3 on the diarrhea scale ranging from 0 (none) to 3 (severe)
Time Frame: At 10 days since enrollment
Population: Participants indicating their adverse effects at 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prone to Diarrhea | Not Prone to Diarrhea
Number analyzed (Participants) | 21 | 105
Participants | 6 | 21

10. Other Pre Specified Outcome: Number of Participants Reporting Severe Diarrhea at Day 10 Among Those Self-identified as Prone or Not Prone to Diarrhea
Description: Among those indicating proneness to diarrhea or not at enrollment, the number who gave a rating of 3 on the diarrhea scale ranging from 0 (none) to 3 (severe)
Time Frame: At 10 days since enrollment
Population: Participants who gave ratings of adverse effects at day 10
Measure: Count of Participants; unit: Participants
Arm/Group | Prone to Diarrhea | Not Prone to Diarrhea
Number analyzed (Participants) | 21 | 80
Participants | 1 | 4

11. Other Pre Specified Outcome: Number of Female Participants Reporting Any Vaginal Symptoms at Day 3 Among Those Self-identified as Prone or Not Prone to Vaginal Itching or Discharge
Description: Female participants contacted after 3 days of treatment were divided into two groups: those who had or had not reported at baseline a proneness to vaginal symptoms. The measure was the number in each group who gave ratings of 1, 2, or 3 on the vaginal symptoms scale, ranging from 0 (none) to 3 (severe), with a higher score indicating more severe symptoms.
Time Frame: After 3 days of treatment
Population: Female participants available at the end of 3 days of treatment who had indicated proneness or not to vaginal symptoms at enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Prone to Vaginal Itching or Discharge: Female participants indicating proneness to vaginal itching or discharge at enrollment
- Not Prone to Vaginal Itching or Discharge: Female participants indicating no proneness to vaginal itching or discharge at enrollment
Arm/Group | Prone to Vaginal Itching or Discharge | Not Prone to Vaginal Itching or Discharge
Number analyzed (Participants) | 24 | 72
Participants | 6 | 11

12. Other Pre Specified Outcome: Number of Female Participants Reporting Severe Vaginal Symptoms at Day 3 Among Those Self-identified as Prone or Not Prone to Vaginal Itching or Discharge
Description: Among female participants indicating a proneness or not to vaginal itching or discharge, the number of ratings of 3 on the vaginal symptom scale ranging from 0 (none) to 3 (severe)Female participants contacted after 3 days of treatment were divided into two groups: those who had or had not reported at baseline a proneness to vaginal symptoms. The measure was the number in each group who gave a rating of 1, 3 on the vaginal symptoms scale, ranging from 0 (none) to 3 (severe), with a higher score indicating more severe symptoms.
Time Frame: At the end of 3 days of treatment
Population: Female participants reporting adverse effects at day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Prone to Vaginal Itching or Discharge | Not Prone to Vaginal Itching or Discharge
Number analyzed (Participants) | 24 | 72
Participants | 0 | 2

13. Other Pre Specified Outcome: Number of Female Participants Reporting Any Vaginal Symptoms at Day 10 Among Those Self-identified as Prone or Not Prone to Vaginal Itching or Discharge
Description: Female participants contacted after 10 days since enrollment were divided into two groups: those who had or had not reported at baseline a proneness to vaginal symptoms. The measure was the number in each group who gave ratings of 1, 2, or 3 on the vaginal symptoms scale, ranging from 0 (none) to 3 (severe), with a higher score indicating more severe symptoms.
Time Frame: At 10 days since enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Prone to Vaginal Itching or Discharge | Not Prone to Vaginal Itching or Discharge
Number analyzed (Participants) | 24 | 53
Participants | 10 | 9

14. Other Pre Specified Outcome: Number of Female Participants Reporting Severe Vaginal Symptoms at Day 10 Among Those Self-identified as Prone or Not Prone to Vaginal Itching or Discharge
Description: Female participants contacted at 10 days since enrollment were divided into two groups: those who had or had not reported at baseline a proneness to vaginal symptoms. The measure was the number in each group who gave rating of 3 on the vaginal symptoms scale, ranging from 0 (none) to 3 (severe), with a higher score indicating more severe symptoms.
Time Frame: At 10 days since enrollment
Population: Female participants giving ratings of adverse effects at day 10
Measure: Count of Participants; unit: Participants
Arm/Group | Prone to Vaginal Itching or Discharge | Not Prone to Vaginal Itching or Discharge
Number analyzed (Participants) | 24 | 53
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 10 days since enrollment
Description: Participants were asked about adverse events at the end of 3 and 10 days. Since they were are office patients, we would have been aware of deaths or serious adverse events
Arm/Group | High Dose | Standard Dose
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/79
Other Adverse Events (participants affected / at risk) | 53/78 | 52/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | High Dose (N=78) | Standard Dose (N=79)
Severe diarrhea at day 3 (Gastrointestinal disorders) | 5/65 (5) | 5/71 (5) — Rating of 3 on a diarrhea scale ranging from 0 (none) to 3 (severe)
Any diarrhea day 3 (Gastrointestinal disorders) | 28/65 (28) | 29/71 (29) — Rating of 1, 2, or 3 on a diarrhea scale ranging from 0 (none) to 3 (severe)
Severe diarrhea day 10 (Gastrointestinal disorders) | 3/49 (3) | 2/58 (2) — Rating of 3 on a diarrhea scale ranging from 0 (none) to 3 (severe)
Any diarrhea day 10 (Gastrointestinal disorders) | 14/49 (14) | 14/58 (14) — Score of 1, 2, or 3 on a diarrhea scale ranging from 0 (none) to 3 (severe)
Severe vaginal itching or discharge day 3 (Infections and infestations) | 2/45 (2) | 0/55 (0) — Rating of 3 on vaginal symptom scale ranging from 0 (none) to 3 (severe)
Any vaginal itching or discharge day 3 (Infections and infestations) | 6/45 (6) | 11/55 (11) — Rating of 1, 2, or 3 on vaginal symptom scale ranging from 0 (none) to 3 (severe)
Severe vaginal discharge or itching day 10 (Infections and infestations) | 1/35 (1) | 0/47 (0) — Score of 3 on vaginal symptoms scale ranging from 0 (none) to 3 (severe)
Any vaginal itching or discharge day 10 (Infections and infestations) | 9/35 (9) | 10/47 (10) — Score of 1, 2, or 3 on vaginal symptom scale ranging from 0 (none) to 3 (severe)

LIMITATIONS AND CAVEATS:
1. Early termination midway in the study after a preliminary analysis demonstrated futility
2. Underestimation of non-serious adverse effects because of dropouts and difficulty contacting participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT03431337/Prot_SAP_000.pdf